CLINICAL TRIAL: NCT03516071
Title: A Multicenter, Randomized, Open-label, Phase II Clinical Study to Evaluate the Efficacy and Safety of Brivanib Alaninate (ZL-2301) Combined With Best Supportive Care (BSC) and Pharmacokinetic Profiles of Brivanib Alaninate in Patients With Advanced Hepatocellular Carcinoma (HCC) Failed or Intolerant of Standard Systemic Chemotherapy and/or Sorafenib
Brief Title: A Phase 2 Study of Brivanib in Chinese Patients With Previously Treated Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZL-2301-001
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular Carcinoma; HCC; Brivanib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — brivanib; BID protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brivanib 800 mg, QD + BSC (Experimental)
  Interventions: Drug: Brivanib 800 mg, QD
- Brivanib 400 mg, BID + BSC (Experimental)
  Interventions: Drug: Brivanib 400 mg, BID

INTERVENTIONS:
Drug: Brivanib 800 mg, QD — Brivanib Alaninate 800 mg QD, PO
  Arms: Brivanib 800 mg, QD + BSC
Drug: Brivanib 400 mg, BID — Brivanib Alaninate 400 mg BID, PO
  Arms: Brivanib 400 mg, BID + BSC

SUMMARY:
This is a Phase 2, Open-label, Randomized, Multicenter Study to Investigate the Efficacy, Safety, and Pharmacokinetics of Brivanib in Patients with Previously Treated Advanced Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years, male or female
* Histologically or cytologically confirmed or the clinical diagnosis standard confirmed hepatocellular carcinoma (HCC) patients
* Failure or intolerance to prior treatment with chemotherapy and/or targeted therapy
* Liver function status Child-Pugh Class A or B (score≤7)
* ECOG Performance Status score 0 or 1
* Patients must have adequate bone marrow, renal and hepatic function

Exclusion Criteria:

* Known history or symptomatic metastatic brain
* Uncontrolled moderate and severe ascites
* With bleeding tendency and thrombosis history
* Known history of severe cardiovascular disease
* Uncontrollable active infections (≥CTCAE Grade 2)
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Disease control rate (DCR) at 3 months from randomization | 12 weeks from randomization
  Defined as the percentage of patients with complete response, partial response, or stable disease at 12 weeks from randomization by RECIST v1.1.
Time to Progress (TTP) | 12 weeks from randomization
  Defined as the time from random assignment to radiologic disease progression.

SECONDARY OUTCOMES:
Disease control rate (DCR) at 6 months from randomization | 24 weeks from randomization
  Defined as the percentage of patients with complete response, partial response, or stable disease at 24 weeks from randomization by RECIST v1.1.
Progression-free survival (PFS) | 24 weeks from randomization
  Defined as the time from random assignment until the date of disease progression or death as a result of any cause.
Objective response rate (ORR) | 24 weeks from randomization
  Defined as the proportion of randomized patients with CR or PR as the optimal response in each treatment group assessed by use of RECIST 1.1 criteria
Overall survival (OS) | 24 weeks from randomization
  Refers to the duration from randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - China PLA 81st hospital, Nanjing, Jiangsu
  - The first Hospital of Jilin University, Changchun, Jilin
  - Army General Hospital of Shenyang military region, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Xi’an, Shanxi
  - West China Hospital West China School of Medicine Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang